CLINICAL TRIAL: NCT00002459
Title: Phase III Randomized Study of Adjuvant Pelvic Radiotherapy Versus Observation Alone in Patients With Completely Resected, Stage I or II, High-Grade Uterine Sarcoma
Brief Title: Radiation Therapy or No Further Treatment Following Surgery in Treating Patients With Cancer of the Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-55874; EORTC-55874; CAN-NCIC-EN4
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Endometrial Cancer; Sarcoma
Keywords: stage I uterine sarcoma; stage II uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Sarcoma; Sarcoma, Endometrial Stromal | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether receiving radiation therapy or no further therapy after surgery is more effective for cancer of the uterus.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with that of no further therapy in treating patients who have stage I or stage II cancer of the uterus that has been surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the rates of pelvic recurrence and development of distant metastases in patients with completely resected, stage I or II, high-grade uterine sarcoma treated with adjuvant pelvic radiotherapy vs observation alone.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, tumor histology (leiomyosarcoma vs mixed mesodermal sarcoma vs endometrial stromal sarcoma), and surgical procedure (total abdominal hysterectomy (TAH) with or without bilateral salpingo-oophorectomy (BSO) vs TAH and BSO with pelvic and para-aortic node sampling and random biopsies). Patients are randomized to 1 of 2 treatment arms. Arm I: Beginning within 6 weeks after surgery, patients undergo pelvic radiotherapy 5 days a week for 5.6 weeks. Arm II: Patients undergo observation alone. Patients are followed every 2 months for 1 year, every 3 months for 2 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 200 patients (100 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven high-grade uterine sarcoma Eligible subtypes: Leiomyosarcoma Mixed mesodermal (mullerian) sarcoma Endometrial sarcoma Surgically proven stage I or II (T1-2, N0, M0) disease No leiomyoma with a high mitotic activity index after hormonal therapy (especially estrogen) Mixoid leiomyosarcoma with a low mitotic activity index allowed Completely resected disease Prior abdominal hysterectomy as minimal surgical procedure required

PATIENT CHARACTERISTICS: Age: Any age Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix No serious mental disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: See Disease Characteristics Radiotherapy: No prior radiotherapy Surgery: See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 1988-04; Primary Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio L. Pecorelli, MD, Study Chair — Spedali Civili di Brescia; Gavin C.E. Stuart, MD, Study Chair — Tom Baker Cancer Centre - Calgary
Locations (28):
- U.Z. Gasthuisberg, Leuven, Belgium
- Canada (2):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
- Centre Henri Becquerel, Rouen, France
- Italy (8):
  - Spedali Civili, Brescia
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Istituto Scientifico H.S. Raffaele, Milan
  - Ospedale San Gerardo, Monza
  - Universita di Padova, Padua
  - I.R.C.C.S. Policlinico San Matteo, Pavia
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale Civile, Voghera (PV)
- Netherlands (9):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Atrium Medical Centre, Heerlen
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - University Hospital - Rotterdam Dijkzigt, Rotterdam
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Medical University of Gdansk, Gdansk, Poland
- Instituto Valenciano De Oncologia, Valencia, Spain
- Sweden (2):
  - University Hospital of Linkoping, Linköping
  - Karolinska Hospital, Stockholm
- Hopital Cantonal Universitaire de Geneva, Geneva, Switzerland
- United Kingdom (2):
  - Derbyshire Royal Infirmary, Derby, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Result] Reed NS, Mangioni C, Malmstrom H, Scarfone G, Poveda A, Pecorelli S, Tateo S, Franchi M, Jobsen JJ, Coens C, Teodorovic I, Vergote I, Vermorken JB; European Organisation for Research and Treatment of Cancer Gynaecological Cancer Group. Phase III randomised study to evaluate the role of adjuvant pelvic radiotherapy in the treatment of uterine sarcomas stages I and II: an European Organisation for Research and Treatment of Cancer Gynaecological Cancer Group Study (protocol 55874). Eur J Cancer. 2008 Apr;44(6):808-18. doi: 10.1016/j.ejca.2008.01.019. Epub 2008 Apr 2. PMID 18378136
- [Result] Reed NS, Mangioni C, Malmstrom H, et al.: First results of a randomised trial comparing radiotherapy versus observation post operatively in patients with uterine sarcomas. An EORTC-GCG study. [Abstract] Int J Gynecol Cancer 13 (Suppl 1): A-PL12, 4, 2003.